CLINICAL TRIAL: NCT07130773
Title: Procedural Comparative Evaluation of Pulmonary Vein Isolation Using the FARAWAVE Nav PFA Catheter Without Pre-Ablation Computer Tomography (CT) vs. Conventional Farapulse With Pre-Ablation CT: A Single Centre Open-label, Randomized Controlled Trial
Brief Title: Comparative Intra-procedural Evaluation of Farapulse and FARAWAVE Nav Catheters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Marco Bergonti, MD PhD, Cardiocentro Ticino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCT2025-FaraRadiation; BASEC-ID 2025-01638 (Other: Swissethics)
Record Dates: First submitted 2025-08-08; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation Ablation; Pulsed Field Ablation
Keywords: pulsed filed ablation; atrial fibrillation; ablation; pulmonary vein isolation; electroanatomical map; ionizing radiation; farapulse; farawave nav
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): FARAWAVE Nav without pre-ablation CT
  Interventions: Device: Second-generation FARAWAVE Nav catheter without the use of pre-ablation CT
- Control (Active Comparator): FARAPULSE with pre-ablation CT
  Interventions: Device: FARAPULSE with pre-ablation CT

INTERVENTIONS:
Device: Second-generation FARAWAVE Nav catheter without the use of pre-ablation CT — FARAWAVE Nav without pre-ablation CT (Intervention Group, n = 29)
  Description of the investigation-specific intervention:
  Participants in the intervention group will undergo pulmonary vein isolation (PVI) using the second-generation FARAWAVE Nav pulsed field ablation (PFA) catheter without the use of pre-ablation CT imaging. The FARAWAVE Nav catheter integrates magnetic navigation and electroanatomical mapping capabilities, allowing real-time visualization of left atrial anatomy and electrical signals. Energy delivery is based on non-thermal pulsed electric fields (irreversible electroporation), specifically targeting myocardial tissue while sparing surrounding structures.
  Arms: Intervention
Device: FARAPULSE with pre-ablation CT — FARAPULSE with pre-ablation CT (Control Group, n = 29)
  Description of the investigation-specific intervention:
  Participants in the control group will undergo pulmonary vein isolation (PVI) using the first-generation FARAPULSE pulsed field ablation (PFA) catheter. All patients in this group will undergo pre-procedural cardiac CT imaging to evaluate pulmonary vein anatomy and assist in procedural planning. The FARAPULSE catheter delivers non-thermal pulsed electric fields for selective myocardial ablation, aiming to achieve electrical isolation of the pulmonary veins.
  Arms: Control

SUMMARY:
The FARAPULSE PFA catheter (Boston Scientific), a first-generation Pulsed Field Ablation (PFA) tool, has demonstrated good performance in isolating pulmonary veins (PV). Several centers, including ours, utilize pre-procedural computer tomography (CT) to evaluate individual pulmonary vein anatomy and optimize ablation planning. However, these imaging modalities are costly. Additionally, CT imaging exposes patients to radiation, and introduce significant logistical challenges to the procedural workflow.

The FARAWAVE Nav PFA catheter, a second-generation device, integrates magnetic navigation capabilities with detailed mapping and PFA therapy into a single tool. This system leverages the FARAVIEW Software Module, offering tailored mapping solutions visualized on the FARAPULSE PFA system, including the creation of voltage and activation maps.

These features address the limitations of the first-generation FARAPULSE catheter and have the potential to improve procedural accuracy and the durability of pulmonary vein isolation. Moreover, they may obviate the need for pre-procedural CT, thereby reducing costs and minimizing patient radiation exposure.

Our study evaluates whether the FARAWAVE Nav catheter, used without pre-ablation CT, allows for a reduction in fluoroscopy time and overall patient radiation exposure compared to the conventional workflow with the FARAPULSE catheter. Furthermore, we will assess procedural time, costs, number of PFA applications, and AF recurrence-free survival

DETAILED DESCRIPTION:
The FARAPULSE PFA catheter (Boston Scientific), a first-generation Pulsed Field Ablation (PFA) tool, has demonstrated good performance in isolating pulmonary veins (PV) as standard of care for atrial fibrillation (AF) ablation. Several centers, including ours, utilize pre-procedural CT or cardiac magnetic resonance (CMR) imaging to evaluate individual pulmonary vein anatomy and optimize ablation planning. However, these imaging modalities are costly. Additionally, CT imaging exposes patients to radiation, and both CT and CMR add significant logistical challenges to the procedural workflow.

The FARAWAVE Nav PFA catheter, a second-generation device, integrates magnetic navigation capabilities with detailed mapping and PFA therapy into a single device. This system leverages the FARAVIEW Software Module, offering tailored mapping solutions visualized on the FARAPULSE PFA System, including the creation of voltage and activation maps. Key technical enhancements of the FARAWAVE Nav PFA catheter include: Field Tag Technology: Field tagging estimates field volume and indicates energy delivery locations. Tags confirm overlap between applications, ensuring comprehensive PV isolation. Voltage/Activation Maps: Mapping data enhances procedure precision, allowing visualization of electrical activation and PV anatomy without reliance on pre-ablation CT imaging. These features address the limitations of the first-generation FARAPULSE catheter and have the potential to enhance procedural accuracy and the durability of pulmonary vein isolation. Moreover, they may eliminate the need for pre-procedural CT or CMR, thereby reducing costs and minimizing patient exposure to radiation.

Our center, like several others, has used the first-generation catheter in routine clinical practice for over a year. More recently, we have also started using the second-generation catheter as part of standard clinical care. Currently, the two devices are used interchangeably, depending on logistical availability, particularly the presence of specialized technicians from Boston Scientific, who are required for the proper operation of the second-generation catheter.

Our study evaluates whether the FARAWAVE Nav catheter, without pre-ablation CT, allows to reduce fluoroscopy time and total patient radiation load as compared to conventional workflow with FARAPULSE catheter. Furthermore, procedural time, costs, number of PFA applications and AF recurrence free survival will be assessed.

Inclusion Criteria

* Atrial fibrillation (AF) documented on a 12-lead ECG, Holter monitor, or implantable cardiac device.
* Candidate for ablation according to current atrial fibrillation guidelines.
* Age ≥18 years at the time of informed consent.
* Signed informed consent obtained.

Exclusion Criteria

* Previous left atrial ablation or left atrial surgery.
* Presence of intracardiac thrombus.
* Persistent atrial fibrillation lasting >3 years.
* Severe mitral regurgitation or moderate-to-severe mitral stenosis.
* Pregnancy (all women under 50 years undergo an HCG blood test prior to inclusion to exclude pregnancy).

Primary Endpoint

1. Fluoroscopy Time (measured in minutes)

Secondary Endpoints 2.1 Total Patient Radiation Load 2.2 Procedural Costs 2.3 Procedure Time 2.4 Left Atrial Dwelling Time 2.5 Fluoroscopy Time After Transseptal Puncture 2.6 Number of PFA Applications 2.7 AF Recurrence-Free Survival 2.8 AF Burden (in Patients with implantable loop recorder) 2.9 AF Burden (All Patients)

Randomization: 58 Patients will be randomized 1:1 to:

1. FARAPULSE + pre-ablation CT (Control Group, n=29).
2. FARAWAVE Nav without pre-ablation CT (Intervention Group, n=29). Randomization will be performed using stratified allocation based on Atrial Fibrillation pattern (paroxysmal vs. persistent AF) in a 1:1 fashion.

Intraprocedural fluoroscopy time will be collected at the time of AF ablation procedure.

To determine the required sample size for this study, we performed calculations based on previous studies, the expected fluoroscopy time are:

Control Group: Mean fluoroscopy time = 12 minutes, SD = 8 minutes [doi.org/10.1161/CIRCULATIONAHA.123.064959] Intervention Group: Mean fluoroscopy time = 7 minutes, SD = 7 minutes [doi:10.1161/CIRCEP.122.011780] Given these assumptions, that correspond to an effect size (Cohen'd) of 0.80, a power of 80% and a 2-sided alpha of 5%, we will need to enrol 52 patients (26 per group). To ensure the study remains adequately powered despite potential dropouts, protocol deviations, or missing data, an additional 10% buffer may be considered, bringing the total recommended enrolment to 58 patients per group. Calculations have been performed using the Stata software (release 18.5, StataCorp, College Station, TX, USA).

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation (AF) documented on a 12-lead ECG, Holter monitor, or implantable cardiac device.
* Candidate for ablation according to current atrial fibrillation guidelines.
* Age ≥18 years at the time of informed consent.
* Signed informed consent obtained

Exclusion Criteria:

* Previous left atrial ablation or left atrial surgery.
* Presence of intracardiac thrombus.
* Persistent atrial fibrillation lasting >3 years.
* Severe mitral regurgitation or moderate-to-severe mitral stenosis.
* Pregnancy (all women under 50 years undergo an HCG blood test prior to inclusion to exclude pregnancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fluoroscopy time | immediately after the procedure
  The primary outcome of this investigation is fluoroscopy time, measured in minutes during the pulmonary vein isolation procedure.
  This outcome was chosen because it directly reflects the amount of radiation exposure experienced by the patient and is a critical measure of procedural efficiency and safety. For patients undergoing PVI plus additional left or right atrial ablations (planned or unplanned) the fluoroscopy time will be counted until the last application of the PVI.
  Fluoroscopic times will be compared between groups using the unpaired Student t test. The mean difference and 95%CI will be computed. In case of skewness, data will be log-transformed before entering the test. In this the mean difference on the log scale and the ratio on the original scale will be presented, both with 95%CI.

SECONDARY OUTCOMES:
Total Patient Radiation Load | immediately after the procedure
  Total patient radiation load (cGy·cm²): to assess overall radiation exposure, including both imaging and intra-procedural sources. In case a patient randomized to the control group has already undergone a cardiac CT scan for another clinical reason in the past, the scan will not be repeated for ethical reasons. However, for the purpose of radiation dose calculation, the average radiation dose of a cardiac CT scan will be added as if the scan had been performed. Conversely, if a patient in the intervention group has previously undergone a cardiac CT scan, the operator will not review this scan prior to the procedure, and the corresponding radiation dose will not be included in the calculation.
  Analysis: same as the primary endpoint
Procedure Time | immediately after the procedure
  Procedure time (minutes): to evaluate procedural efficiency from catheter insertion to removal. For patients undergoing PVI plus additional left or right atrial ablations (planned or unplanned) the procedure time will be counted until the last application of the PVI.
  Analysis: same as the primary endpoint
Left Atrial Dwelling Time | immediately after the procedure
  Left atrial dwelling time (minutes): to assess the duration of catheter presence in the left atrium, which is associated with thromboembolic and procedural risks.
  Analysis: same as the primary endpoint.
Fluoroscopy Time After Transseptal Puncture | immediately after the procedure
  Fluoroscopy time after transseptal puncture (minutes): to determine radiation exposure specifically during the left atrial portion of the procedure.
Number of PFA Applications | immediately after the procedure
  Number of PFA applications: to evaluate treatment burden and procedural complexity.
AF Recurrence-Free Survival | up to 6 months
  AF Recurrence-Free Survival: Freedom from AF, atrial flutter, or atrial tachycardia lasting >30 seconds, documented by ILR, over a 12-month follow-up, after two months of blanking period. Kaplan Meier event-free curves will be presented for each group and compared with the logrank test. Hazard ratios (HR) and 95%CI will be derived from a Cox model. Follow-up will start after the two months blanking period. Patients who die without atrial arrhythmia recurrence will be censored at the time of death
AF Burden | up to 6 months
  AF Burden: Proportion of time in AF, as assessed by the ILR over 6 months or 7 days Holter monitor. The same analysis as for the primary endpoint will be used.

OTHER OUTCOMES:
Procedural Costs | immediately after the procedure
  Procedural costs: Pre-procedural imaging and procedural costs [Cost of CT scan, FARAPULSE Catheter, FARAVEIW Catheter.] The same analysis as for the primary endpoint will be used. In addition the ICER - incremental cost-effectiveness ratio - will be computes as the ratio of the difference in costs over the difference in effect as measures for the primary endpoint

IPD SHARING:
Plan to Share IPD: No